CLINICAL TRIAL: NCT00459420
Title: Caffeine for Excessive Daytime Somnolence in Parkinson's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ron Postuma (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Ron Postuma, Neurologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN-06-68
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease; Excessive Daytime Somnolence
Keywords: Parkinson's disease; Excessive Daytime Somnolence; Caffeine; Disease-Modifying
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence | interventions — Caffeine; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Caffeine (Experimental)
  Interventions: Drug: Caffeine 100-200 mg BID

INTERVENTIONS:
Drug: Caffeine 100-200 mg BID — Caffeine 100 mg BID for three weeks, then 200 mg BID for three weeks, then 100 mg BID for 1 week, then placebo
  Arms: Caffeine
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
Many patients with Parkinson's disease (PD) have sleep problems, including excessive sleepiness during the day. This is probably due to degeneration of sleep-regulating areas in the brain. At present, the only treatment for sleepiness in PD is modafinil, which is expensive and only partially effective. There is another potential treatment for sleepiness that is used worldwide, is inexpensive, well tolerated and safe - namely, caffeine. There have also been suggestions that caffeine may slow the progression of degeneration in PD, since coffee non-drinkers are at higher risk of developing PD. PD patients, even with severe sleepiness often do not use caffeine. It is unclear whether this is because their PD makes their sleepiness unresponsive to caffeine, because they cannot tolerate it, or whether this reflects their lifelong habit of non-use. This proposal outlines a trial in which patients with excessive sleepiness will be given caffeine or placebo (no therapy) in a blinded fashion. In this way, the effect of caffeine on sleepiness and motor symptoms can be directly analyzed. In addition, these findings can be used to test the tolerability of caffeine, to help plan a larger-scale study testing whether caffeine can slow the progression of PD

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disorder characterized by motor disability and many disabling non-motor symptoms. Excessive daytime somnolence (EDS) is found in up to 50% of patients with PD, and can cause considerable impairment of quality of life. At present, the only proven treatment for EDS in PD is modafinil, an alerting agent with an unknown mechanism of action. However, modafinil is only moderately effective and is very expensive. Caffeine is a very well tolerated and inexpensive alerting agent that is used worldwide, but very few patients with PD use it as therapy for EDS. It is unclear whether this is because it does not help EDS in PD, has side effects, or simply has not been considered because of lifelong patterns of non-use.

If caffeine can be demonstrated as an effective agent for EDS in PD, it will likely become the first-line agent for EDS. This will result in considerable cost savings for patients and health care payers, as well as potentially helping those who cannot tolerate, do not respond to, or cannot afford modafinil.

Another compelling question of interest to patients with PD is whether caffeine may be neuroprotective. Despite intensive research, no treatment has been found that can slow the progression of neurodegeneration in PD. Recently numerous epidemiologic studies have linked lifelong use of caffeine to a lower risk of PD. Although the mechanism for this finding is unclear, supporting evidence from animal models suggests that a true neuroprotective benefit of caffeine is a strong possibility. Alternatively, caffeine could have a benefit on motor manifestations of PD, which would prevent diagnosis of PD. Any finding of a symptomatic benefit of caffeine on motor manifestations of PD will have obvious and important implications for treatment of persons affected with PD and for planning of neuroprotective trials. Any finding of a neuroprotective benefit of caffeine will almost certainly result in its immediate widespread use in PD, with profound implications for patient care.

The present proposal is for a double blind randomized placebo controlled crossover trial that will answer three important questions in PD: is caffeine useful for the treatment of EDS in patients with PD? does caffeine have any symptomatic effect on the motor manifestations of PD? and, does caffeine have an acceptable tolerability and side effect profile that will allow planning of an eventual neuroprotective trial? Patients with PD who have EDS with an Epworth sleepiness scale of >10 will be randomized to caffeine therapy (100 mg twice per day for three weeks, then 200 mg twice per day for three weeks) or placebo. A final assessment will be performed after a 4-week washout. A total of 52 patients will be randomized over a two-year period. The primary outcome measure will be the change in Epworth sleepiness scale between patients receiving caffeine versus placebo. Secondary outcome measures will include other sleep scales, tolerability measures, and measures of motor function and overall quality of life. After tests to assess normal distribution, analysis will be with two-sample t-test.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic PD
* Excessive daytime somnolence (defined as an Epworth sleepiness scale score of >10).

Exclusion Criteria:

* Estimated daily caffeine intake of more than 200 mg per day
* Active peptic ulcer disease
* Supraventricular cardiac arrhythmia (such as atrial fibrillation or atrial flutter)
* Uncontrolled hypertension - defined as systolic bp >170 or diastolic bp >110 on two consecutive readings
* EDS is caused by sleep apnea, restless legs syndrome, narcolepsy, shift work, or sleep promoting agents.
* Current use of prescribed alerting agents such as modafinil and methylphenidate
* Pre-menopausal women who are not using effective methods of birth control
* Dementia, defined as MMSE <24/30 and ADL impairment secondary to cognitive loss, or inability to understand consent process
* Depression, as defined by a Beck Depression Inventory score of >15.
* Changes to antiparkinsonian medication in the last 3 months, or changes to antiparkinsonian medication are anticipated during the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in Epworth Sleepiness Scale | 3 weeks

SECONDARY OUTCOMES:
Unified Parkinson Disease Rating Scale | 3 weeks
Clinical Global Impression of Change | 3 weeks
Pittsburgh Sleep Quality Index | 3 weeks
Fatigue Severity Scale | 3 weeks
Stanford Sleep Scale | 3 weeks
PDQ-39 | 3 weeks
SF-36 | 3 weeks
Tolerability of Caffeine | 3 weeks
Beck Depression Inventory | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ron Postuma, MD, MSc, Principal Investigator — Montreal General Hospital
Locations (2):
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec